CLINICAL TRIAL: NCT03050996
Title: Intraoperative Evaluation or Retrograde Leack Point Pressure During Robot Assisted Radical Prostatectomy for Proper Autologous Suburethral Sling Tensioning to Improve Early Urinary Continence Recovery
Brief Title: Retrograde Perfusion Sphinterometry and Autologous Sling to Improve Urinary Continence in Robotic Radical Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, acestari, Head Department of Urology, Istituto Auxologico Italiano
Other Study IDs: IAI-URO-RPS-RALP
Record Dates: First submitted 2017-02-05; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- robotic radical prostatectomy patients: Patient scheduled to undergo robotic assisted radical prostatectomy
  Interventions: Procedure: robotic radical prostatectomy

INTERVENTIONS:
Procedure: robotic radical prostatectomy — Urodynamic evaluation during robotic radical prostatectomy
  Other Names: Questionnaires

SUMMARY:
Urinary continence recovery remains one of the most bothersome side effect of modern radical prostate surgery and several technical modifications, especially in Robotic assisted radical prostatectomy procedures, have been reported in order to improve early urinary continence recovery.

With the aim to improve the urinary continence recovery after robotic prostatectomy, we evaluate the impact of the use of a 6-branch retropubic suburethral autologous sling, created and placed during the procedure, in association with intraoperative evaluation of the retrograde leak point pressure by means of retrograde perfusion sphincterometry for proper sling tensioning.

DETAILED DESCRIPTION:
Retrograde leak point pressure (RLPP) is intraoperatively evaluated, by means of retrograde perfusion sphinterometry, in patients scheduled to undergo RALP at our Institution, with no patient affected by preoperative urinary incontinence or neurological disorders.

Retrograde Perfusion Sphincterometry (RPS) technique. With the patient under general anaesthesia, with a nasogastric tube and rectal tube to decompress the bowel, properly positioned for RALP procedure (30° of trendelemburg), a graduated fluid supporting pole is positioned in order that the 0 cm position resulted at the level of patient's pubis . At the beginning of the surgical procedure, the indwelling 16ch Foley catheter is inserted and the bladder fully emptied.

The deflated Foley catheter is then retracted to mid urethra/fossa navicularis and inflated with 1.5 cc of Saline in order to prevent fluid extravasation from the external meatus. The catheter is then connected to a 500 cc of Saline perfusate bottle and the bottle is progressively lowered (along the fluid supporting pole) from an eight of 1 meter above the pubis till the fluid stops to flow. The value, in cmH2O, at which the fluid stops to flow into the bladder represents the RLPP.

Six-branch autologous sling surgical technique. Briefly, after bilateral vas deferens harvesting at the time of bladder mobilization during RALP, the sling is prepared on scrub nurse table with six absorbable CT2 needle 0-Vicryl sutures (each measuring 16 cm in length), tight centrally together; the vas deferens are cut in 6 specimens and transfixed with the suture and collected centrally in order to create the bulky central part of the sling .

Before urinary continuity restoration, the sling is introduced into the surgical field and its extremities are fixed bilaterally to the periosteum of the pubic branches at medial (just lateral to the symphysis), lateral and posterior level; the denonvilliers fascia is restored in a double layer fashion in order to separate the urethrovesical anastomosis from the sling. Upon completion of the urethrovesical anastomosis, the sling is tensioned, tightening together the two medial branches first, then the two lateral ones. After subjective proper tension is achieved, the RLPP is evaluated and the tension adjusted accordingly to pre surgery values.

RLPP was respectively evaluated before pneumoperitoneum induction (RLPPb) and after pneumoperitoneum induction (RLPPp). RLPP was then evaluated after urethrovesical anastomosis (RLPPa) and during proper sling tensioning (RLPPs). The aim of sling tensioning was to obtain similar pressures as after pneumoperitoneum induction (RLPPs ≅RLPPp).

ELIGIBILITY:
Inclusion Criteria:

* Hystopathologically confirmed prostate cancer

Exclusion Criteria:

* Preoperative urinary incontinence
* Neurological disorders

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient affected by prostate cancer, scheduled to undergo robotic assisted radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-05-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Impact of radical prostatectomy and autologous suburethral placement on sphincteric apparatus and early urinary continence recovery | Intraoperative evaluation of sphincteric efficacy with Retrograde Leak Point Pressure evaluation - post operative recovery of urinary continence at catheter removal - 10 and 30 days after catheter removal - 6 and 12 months after surgery
  evaluation of sphincteric competence after prostate ablation and sling placement under urodynamic evaluation (Retrograde Leak Point Pressure in cmH2O) and recovery of urinary continence (number of pads used)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cestari, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Andrea Cestari, Milan, Italy

IPD SHARING:
Plan to Share IPD: No